CLINICAL TRIAL: NCT07134452
Title: Comparison of Isokinetic Muscle Strength, Grip Strength, Weight Bearing, Proprioceptive Sense, Reaction Time and Functional Parameters Between Subjects With Scapholunate Instability and Healthy Individuals: A Cross-sectional Study
Brief Title: Comparison of Strength, Weight Bearing, Proprioception, Reaction Time and Function in Scapholunate Instability
Status: Active, not recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Principal Investigator, Arzu Dağ, Doctorate student, Hacettepe University
Other Study IDs: 2025/659
Record Dates: First submitted 2025-08-11; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Scapholunate Interosseous Ligament Injury; Scaphoid-Lunate Instability; Scapholunate Dissociation
Keywords: Scapholunate Instability; Isokinetic Muscle Strength; Weight Bearing; Proprioceptive Sensation; Reaction Time; Functionality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scapholunate Instability Group: Individuals diagnosed with scapholunate interosseous ligament injury confirmed by clinical and radiological assessment. Participants will undergo baseline evaluations including isokinetic muscle strength, grip strength, weight-bearing capacity, proprioception, reaction time, and functional assessments.
  Interventions: Diagnostic Test: Baseline Assessments
- Healty Controls: Age- and sex-matched healthy individuals with no history of wrist injury or upper extremity musculoskeletal disorders. Participants will undergo the same baseline evaluations as the scapholunate instability group.
  Interventions: Diagnostic Test: Baseline Assessments

INTERVENTIONS:
Diagnostic Test: Baseline Assessments — Evaluation of isokinetic muscle strength, grip strength, upper extremity weight-bearing capacity, proprioceptive sense, reaction time, and functional performance in both groups

SUMMARY:
Scapholunate (SL) instability is the most common type of instability seen in the wrist, resulting from SLI injury or excessive mobility [1,2]. It usually occurs after trauma and can range from mild injury to severe malalignment [3]. Symptoms include dorsal pain, clicking sound, limited movement, increased pain with weight-bearing, and weakness [4,5]. Pain reduces joint movement and grip strength, limiting daily activities [6]. If there is no dislocation, conservative treatment (education, exercise, splinting) is applied [7].

The wrist absorbs and transfers load through ligaments. During flexion-extension, the scaphoid and lunate follow the capitate [10]. SLIL injuries alter forearm muscle activation. EKRL, EKRB, APL, and FKR are "scapholunate-friendly" muscles; EKU is not recommended due to its pronator effect [12-15]. SLIL mechanoreceptors enhance dynamic stability [11,19]. There are no studies objectively measuring the strength of these muscles.

Isokinetic muscle assessment has not been performed in SL instability. These measurements objectively determine muscle strength and imbalances, personalizing treatment. Weight transfer capacity, reaction time, and proprioception have also not been studied. However, weight transfer is an indicator of stability, proprioception is critical for functionality, and reaction time reflects neuromuscular response speed [23-27].

The aim of this study is to compare forearm isokinetic muscle strength, grip strength, weight transfer, proprioception, reaction time, and functionality in individuals with SL instability with those in healthy individuals.

DETAILED DESCRIPTION:
Scapholunate (SL) instability is the most common type of instability in the wrist, resulting from injury or excessive mobility of the scapholunate interosseous ligaments (SLIL) [1,2]. This condition, which typically arises following trauma, can range in severity from partial ligament injury to irreparable ligament damage and malalignment [3]. Symptoms include dorsal pain, clicking sounds, limited range of motion, a sensation of catching, pain exacerbated by loading, and weakness [4,5]. Pain that occurs during weight-bearing can reduce joint range of motion and grip strength, thereby limiting daily living activities [6]. In cases without radiological findings of dislocation, conservative treatment (education, exercise, splinting) is preferred [7].

The wrist facilitates load absorption and transfer through complex mechanisms and ligaments. During flexion and extension, the scaphoid and lunate follow the movement of the capitate [10]. In SLI injuries, impaired ligament-muscular reflexes alter the activation patterns of the forearm muscles. Among these muscles, the extensor carpi radialis longus (ECRL), extensor carpi radialis brevis (ECRB), abductor pollicis longus (APL), and flexor carpi radialis (FCR) are defined as scapholunate-friendly; the extensor carpi ulnaris (ECU) has been reported as a muscle to be avoided due to its intracarpal pronator effect [12-15].

In recent years, it has been emphasized that static stability approaches are insufficient and that neuromuscular control has gained importance [2]. It has been shown that the SLIL and wrist ligaments are rich in mechanoreceptors and that these structures increase dynamic stability by activating the forearm muscles [11,19]. However, there are no studies that objectively measure the strength of the scapholunate-friendly muscles.

There is no information in the literature regarding the evaluation of wrist muscles in SL instability using an isokinetic system. Isokinetic measurements are also extremely limited in other pathologies affecting the wrist [20-22]. Isokinetic devices measure muscle strength at a constant speed, objectively determining performance at different speeds and revealing muscle imbalances. This enables treatment plans to be personalized.

Similarly, there are no studies examining parameters such as weight transfer capacity, reaction time, and proprioception in SL instability. However, upper extremity load transfer is an important indicator of stability [23-25], and proprioception is critical for functionality. Reaction time indicates the neuromuscular system's ability to respond quickly, and it is thought that this mechanism may be affected in instability [26,27].

This study aims to investigate forearm isokinetic muscle strength, grip strength, weight transfer capacity, proprioceptive sensation, reaction time, and functionality in individuals with scapholunate instability compared to healthy individuals.

Hypotheses H1: Isokinetic forearm muscle strength in patients with SL instability differs from that in healthy individuals.

H2: Grip strength differs between patients with SL instability and healthy individuals.

H3: Proprioceptive sensation differs between patients with SL instability and healthy individuals.

H4: Reaction time differs between patients with SL instability and healthy individuals.

H5: Weight transfer onto the hand differs between patients with SL instability and healthy individuals.

H6: Upper extremity functionality differs between patients with SL instability and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Applying to the clinic within the last 6 months
* Being diagnosed with dynamic scapholunate instability

Exclusion Criteria:

* Having a history of previous hand or wrist surgery,
* Having a history of Reflex Sympathetic Dystrophy,
* Having a Scapholunate Advanced Collapse lesion,
* Having a serious systemic neurological, or psychiatric illness,
* Having been undergoing upper extremity rehabilitation in the last six months, did not wish to participate in the study, or were unable to follow the protocols.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18-45 years. The case group will include individuals diagnosed with scapholunate instability confirmed by clinical and radiological examination. The control group will consist of age- and sex-matched healthy individuals with no history of wrist injury or upper extremity musculoskeletal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic Muscle Strength Evaluation | Baseline
  It will be evaluated with the Isokinetic Cybex device. At 60/90/ angular velocities, the extensor-flexor peak torque force / work produced by the muscle will be evaluated concentrically.
Weight-Bearing Test | Baseline
  Test protocol: The subject will be asked to apply as much pressure as possible with the extended elbow and wrist on a digital scale. The subjects will perform 3 trials and the average value will be recorded in kilograms and will be compared with the weight transfer test of the unaffected hand, which is determined as a normative value for maximum weight-bearing capacity.
Grip Strength Evaluation | Baseline
  It will be evaluated with the JAMAR hand held dynamometer
Wrist Proprioception Evaluation | Baseline
  t will be evaluated with the Isokinetic Cybex Device device The hand will be brought to the target angle value of 30 degrees extension or 30 degrees flexion with the help of a physiotherapist and will be waited for approximately 5 seconds. After the patient learns, he/she will be asked to do it himself/herself with his/her eyes closed. After the movement is repeated 3 times in a row, the participant will be asked to actively apply the determined target extension movement to the same extremity. The difference between the target angle and the measured angle.The difference between the target angle and the measured angle will be recorded as the margin of error.
Reaction Time Evaluation | Baseline
  Upper extremity reaction time evaluation will be performed with the reaction speed measurement and exercise set Blazepod Trainer (Blazepod Trainer Device, Play Coyotta Ltd. Tel Aviv Israel) device. Individuals will be asked to turn off the 5 LEDs placed on the table in front of them as quickly as possible with one hand in the sitting position. Both hands will be evaluated. The number of LEDs extinguished in 30 seconds (number), the unit extinguishing time (msec) and the number of LEDs missed when the LEDs extinguished after a 5-second waiting period will be recorded. Measurements will be made on both hands.
Pain Evaluation | Baseline
  It contains 10 cm line that should be assigned according to perceived pain intensity at rest, during activity and while exercising.
Quick DASH | Baseline
  The QuickDASH is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.

SECONDARY OUTCOMES:
PRWHE (Patient-Rated Wrist/Hand Evaluation) | Baseline
  Patient-Rated Wrist/Hand Evaluation (PRWHE) is a self-reported questionnaire designed to assess wrist and hand pain and functional status. It consists of 15 items, including 5 pain-related questions and 10 function-related questions. Each item is scored on a 0-10 scale, with higher scores indicating greater pain or disability. The total score ranges from 0 (best) to 100 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Dağ, Principal Investigator — Hacettepe University
Locations (1):
- Istanbul Yeni Yuzyil University, Istanbul, Cevizlibag / Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No